CLINICAL TRIAL: NCT05735769
Title: Gender-dependent Symptoms Following Anti-COVID-19 Vaccine in a Lebanese and Italian Populations
Brief Title: Anti-COVID-19 Vaccine Side Effects
Acronym: VAX-IT-LEB
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Collaborators: Lebanese University (Other)
Responsible Party: Principal Investigator, piero portincasa, Professor, MD, University of Bari
Other Study IDs: VaxITLB-19 2021
Record Dates: First submitted 2023-02-17; First posted 2023-02-21 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Vaccine Adverse Reaction; Gender; COVID-19 Vaccine Adverse Reaction
MeSH Terms: conditions — Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2021 and following the COVID-19 (corona virus disease 2019) pandemic, different vaccines were initially authorized in Italy and Lebanon. Notably, vaccine side effects were poorly recorded. Thus, the investigator performed a survey study to monitor COVID-19 vaccine side effects among Italian and Lebanese citizens according to gender and age through a web-based questionnaire in Italian and Arabic languages including 21 items by "Google Form", investigating 13 symptoms, and employing social-media platforms

DETAILED DESCRIPTION:
The COVID-19 pandemic has presented a real challenge to the public health system worldwide since the year 2019, spreading to more than 200 countries and regions worldwide.The emergence and rapid spread of COVID-19 were caused by the coronavirus SARS-CoV-2. Worldwide, the use of COVID-19 vaccines was initially authorized for emergency use and the side effects were not stated clearly. Common side effects were expected but specific side effects linked with COVID-19 vaccines remained uncertain. In this context, survey studies are needed for a comprehensive evaluation of the relationships between vaccine administration, related undesired effects and vaccine safety.

This study represents the first survey following early COVID-19 vaccines administration in two geographic areas, comparatively considering possible differences due to gender and age. A web-based survey was conducted on a cohort of 1975 Italian and 822 Lebanese people who received at least one dose of COVID-19 vaccine. The study was conducted between March and July 2021 on a voluntary basis, and by a tailored anonymous web-based questionnaire. The protocol was approved by the local Ethics Committee, University of Bari 'Aldo Moro' (study number 6752, protocol number 0031044). A specific questionnaire was designed in English and translated into Italian and Arabic. It contains 21 items including demographic data, the history of vaccine administration before COVID-19, the administration of the first and second dose of COVID-19 vaccine, and possible adverse effects.

The survey link was shared by a "Google Form" employing social-media platforms or by personal interview.

The questionnaire explored the presence of 13 possible symptoms appearing following the administration of the first and second dose of COVID-19 vaccine: pain at the injection site, redness at the injection site, swelling at the injection site, induration at the injection site, allergic-urticarial reaction, anaphylaxis, fever (>37 °C), diarrhea, vomiting, asthenia/fatigue, muscle pain, rash, sleepiness/insomnia, irritability/nervousness, headache, lymphadenopathy. The presence and intensity of symptoms were assessed semi-quantitatively by a Visual Analogue Scale (VAS). Besides symptoms, the following aspects were also evaluated: need of drug intake, consultation of a doctor, emergency admission to hospital, and possible hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Anti-COVID-19 vaccine

Exclusion Criteria:

* Subjects who living outside Italy or Lebanon

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Random sample from the Italian and Lebanese population who received first or first and second dose of anti-COVID-19 vaccine
Sampling Method: Non-Probability Sample
Enrollment: 2797 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Symptoms post anti-COVID-19 vaccine | 5 months
  The questionnaire explored the presence of 13 possible symptoms appearing following the administration of the first and second dose of COVID-19 vaccine: pain at the injection site, redness at the injection site, swelling at the injection site, induration at the injection site, allergic-urticarial reaction, anaphylaxis, fever (>37 °C), diarrhea, vomiting, asthenia/fatigue, muscle pain, rash, sleepiness/insomnia, irritability/nervousness, headache, and lymphadenopathy

SECONDARY OUTCOMES:
Severity score post-vaccine anti-COVID-19 | 5 months
  The severity score of symptoms was calculated as follows: [∑ (symptom * duration in hrs * intensity in VAS (visual analog score)] + use of antipyretic drugs (1point) + use of other analgesic drugs (1 point) + recourse to a doctor (1 point) + recourse to emergency room without admission to the ward (1 point) + admission to hospital ward (1 point). The range of the severity score was from 0 to 216 after first dose or second dose

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Sciences and Human Oncology - Clinica medica "A. Murri", Bari, BA, Italy